CLINICAL TRIAL: NCT00021021
Title: A Phase II, Open-Label, Multicenter Trial of Angiozyme in Subjects With Metastatic Renal Cell Cancer
Brief Title: RPI.4610 in Treating Patients With Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ribozyome (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068739; UCLA-001201501; RPI-0004; NCI-G01-1975
Record Dates: First submitted 2001-07-11; First posted 2004-02-16 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2002-05

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; clear cell renal cell carcinoma
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Angiozyme

INTERVENTIONS:
Biological: anti-FLT-1 ribozyme

SUMMARY:
RATIONALE: RPI.4610 may stop the growth of metastatic kidney cancer by stopping blood flow to the tumor.

PURPOSE: Phase II trial to study the effectiveness of RPI.4610 in treating patients who have metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate of patients with metastatic renal cell cancer treated with RPI.4610. II. Determine the percentage of these patients with stable disease at 16 weeks after starting treatment with this drug. III. Assess the safety and tolerability of this drug in these patients.

OUTLINE: This is a multicenter study. Patients receive RPI.4610 subcutaneously daily. Treatment continues for 16 weeks in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease may continue treatment after 16 weeks. Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed clear cell renal cell cancer Stage IV Measurable disease Bone metastases may not be only measurable lesions Failed prior interleukin-2 (IL-2) therapy (with or without interferon) or ineligible or intolerant of IL-2 Prior nephrectomy (radical, partial, or laparoscopic) at least 4 weeks ago No CNS metastases on CT scan or MRI of head

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Hemoglobin greater than 9.5 g/dL No history of bleeding disorder Hepatic: AST or ALT no greater than 3 times upper limit of normal (ULN) Bilirubin no greater than 1.5 times ULN (unless history of Gilbert's syndrome) Alkaline phosphatase no greater than 2.5 times ULN PT no greater than 15 sec INR no greater than 1.5 No history of cirrhosis Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No New York Heart Association class III or IV heart disease No uncontrolled hypertension, defined as newly diagnosed but untreated or treated but with diastolic blood pressure at least 95 mmHg or systolic blood pressure at least 160 mmHg Other: HIV negative No systemic infection requiring antibiotics within the past 28 days No other malignancy within the past 5 years except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix No alcohol or drug abuse within the past 2 years No other medical or psychiatric condition that would preclude study Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 1 month after study

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics At least 4 weeks since prior IL-2 At least 6 months since prior biotherapy for metastases (e.g., vaccines, matrix metalloproteinase inhibitors, or antibody therapy) No prior antiangiogenic agent, including thalidomide, or experimental antiangiogenic agents No concurrent immunotherapy No other concurrent biotherapy Chemotherapy: No prior chemotherapy for metastatic renal cell cancer No concurrent chemotherapy Endocrine therapy: No concurrent estrogens or other hormonal therapy including androgens Concurrent replacement doses of steroids allowed provided stable for the past 28 doses Radiotherapy: At least 8 weeks since prior radiotherapy No concurrent radiotherapy Surgery: See Disease Characteristics At least 4 weeks since prior major surgery Other: At least 4 weeks since prior investigational drugs No other concurrent investigational drugs No concurrent immunosuppressive medications No concurrent warfarin, heparin, low molecular weight heparin, or other anticoagulant agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-09; Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Figlin, MD, FACP, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States